CLINICAL TRIAL: NCT05559450
Title: A Multicenter ,Prospective, Randomized Clinical Trial of Blinatumomab As a Bridge to Allogeneic Hematopoietic Stem Cell Transplantation in High Risk Precursor B-cell Acute Lymphoblastic Leukemia
Brief Title: Blinatumomab as a Bridge to Allo-HSCT in HR BCP-ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Zhongda Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First People's Hospital of Changzhou (Other); Wuxi People's Hospital (Other); First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Principal Investigator, HAN Yue, Director, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022019
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2021-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Blinatumomab arm (Experimental): On the 1st to 3rd day, Blinatumomab should be continuous intravenous use for 24 hours with 9ug/ day for those whose weight are equal to or greater than 45kg, and 5ug/ m2 / day for those whose weight are less than 45kg (maximum dosage is 9ug/ day) per 24 hours. On the 4th to 14th day, for the patients who are equal to or greater than 45kg, they will receive Blinatumomab at the dose of 28ug/ day with continuous intravenous administration, and those below 45kg are given a 24h continuous infusion of 15ug/ m2 / day (maximum dose is 28ug/ day). Bucy-based myeloablative conditioning regimen will be performed on the 15th day.
  Interventions: Drug: Blinatumomab
- Conventional therapy (Other): Bucy-based myeloablative conditioning regimen will be given to those patients are enrolled into control group.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be bridged to conventional BUCY conditioning regimen.
  Arms: Blinatumomab arm
Other: Conventional therapy — Control group will be given conventional BUCY conditioning regimen.
  Arms: Conventional therapy

SUMMARY:
To explore the efficacy and safty of Blinatumomab as a bridge to Allogeneic Hematopoietic Stem Cell Transplantation in High Risk Precursor B-cell Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
High Risk Precursor B-cell Acute Lymphoblastic Leukemia is a kind of leukemia with poor prognosis. Here, we want to explore the efficacy and safty of Blinatumomab as a bridge to Allogeneic Hematopoietic Stem Cell Transplantation in High Risk Precursor B-cell Acute Lymphoblastic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. The patients meet the diagnostic criteria for high risk precursor B-ALL (according to the 2016 WHO classification) and are under hematologic remission.
2. ECOG score is 0-2.
3. Expecting life span is more than 6 months.
4. Patients are free from severe organ dysfunction.

Exclusion Criteria:

1. Patients are combined with severe organ dysfunction: Organ failure: Cardiac failure: ejection fraction(EF) <30%, NYHA standard, cardiac function not Full Grade II or above; Liver and kidney insufficiency: serum total bile Erythroid ≥2mg/dl, AST or ALT≥ upper limit of normal 2.5-fold, serum creatinine (SCr) >2.5mg/ dL or blood Creatinine clearance rate < 30ml/min.
2. Patients are combined with infection or other complications that can not tolerate chemotherapy.
3. Patients are suffering from central nervous system/solitary extramedullary leukemia.
4. Patients are considered as tumer progression.
5. Patients has undergone allogeneic hematopoietic stem cell transplantation or underwent autologous stem cell transplantation within 6 weeks or other immunotherapy within 4 weeks.
6. Pregnant and lactating women will not be included.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the 1st day to the 720th days after enrollment.
  The time from randomization to death from any cause.

SECONDARY OUTCOMES:
The proportion of patients with negative minimal residual disease (MRD) | From the 1st day to the 720th days after enrollment.
  Negative MRD is defined as below 10-4 by flow cytometry.
Progression-Free Survival (PFS) | From the 1st day to the 720th days after enrollment.
  It is defined as the total survival of a patient after the hematopoietic stem cell transplantation, until the tumor recurrence or death from any cause.
Cumulative incidence of relapse (CIR) | From the 1st day to the 720th days after enrollment.
  From hematopoietic stem cell transplantation to recurrence, relapse-free death was considered a competing risk event.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, MD/PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The first affiliated hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182

DOCUMENTS (1):
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT05559450/ICF_000.pdf